CLINICAL TRIAL: NCT05769621
Title: A Retrospective Cohort Study to Characterize Propionic Acidemia Patients
Brief Title: A Retrospective Study to Characterize Participants With Propionic Acidemia
Status: Recruiting | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-3927-P002
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Propionic Acidemia
MeSH Terms: conditions — Propionic Acidemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PA Participants: Participants with PA who meet all eligibility criteria for medical record abstraction.

SUMMARY:
This is a non-interventional, observational, global, multicenter, study describing participant characteristics, clinical outcomes, and event rates in participants with propionic acidemia (PA).

DETAILED DESCRIPTION:
Data will be abstracted through medical record review ensuring inclusion only of data from participants meeting all the inclusion criteria and none of the censoring criteria. Data will be collected retrospectively from study sites, including medical clinics, hospitals and academic medical centers.

ELIGIBILITY:
Inclusion Criteria:

Participants' medical records are eligible for abstraction only if all of the following criteria apply:

* Confirmed diagnosis of PA based on diagnosis by molecular genetic testing (propionyl-CoA carboxylase subunitα[PCCA] and/or propionyl-CoA carboxylase subunitβ[PCCB] mutations).
* Participant provided informed consent (and assent, as applicable).
* Medical records with sufficient data to support medical encounter for CEC adjudication (MEA adjudication) must be available dating back to birth or 01 January 2015, whichever occurs later. Participants born prior to 2015 will require additional information to confirm eligibility.
* Experienced at least one MDE in the 24 months preceding the Index Date or experienced at least 3 MDEs within any one 12-month retrospective review period (based on Index Date) dating back to birth or 01 January 2015, whichever occurs later.
* Must have a confirmed age (months) of disease onset (early or late, where early is defined as the neonatal period).
* Participants who meet any of the censoring criteria listed below may be enrolled into the study if they have a minimum of 2 years of data available for abstraction prior to meeting the censoring criteria and they meet all inclusion criteria based on the data available for abstraction.

Censoring Criteria:

Participants medical records meeting the following censoring criterion will not be abstracted:

* Participation in a clinical study of any investigational agent.
* Received gene therapy treatment
* Confirmed organ transplantation
* Investigator is no longer able to obtain relevant clinical information of the participant.
* Death

Exclusion Criteria:

Participant's medical records will not be eligible for abstraction if the participant meets the following exclusion criteria:

- Participation (prior or ongoing) in clinical study mRNA-3927-P101 (NCT04159103) or mRNA-3927-P101-EXT (NCT05130437).

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals of a minimum age of 2 years with confirmed diagnosis of PA.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Annualized Clinical Event Committee (CEC)-adjudicated Metabolic Decompensation Events (MDEs) | Up to 10 years

SECONDARY OUTCOMES:
Number of CEC-adjudicated MDEs as Assessed by a Pre-Specified Severity Rating Scale | Up to 10 years
Number of Annualized CEC-adjudicated PA-related Hospitalizations | Up to 10 years
Number of Annualized CEC-adjudicated MDE-related Hospitalizations | Up to 10 years
Number of Annualized CEC-adjudicated PA-related Urgent Healthcare Visits | Up to 10 years

CONTACTS AND LOCATIONS:
Locations (29):
- United States (6):
  - University of Stanford Medical Center, Stanford, California
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Royal Children's Hospital Melbourne, Parkville, Victoria, Australia
- Stollery Children's Hospital University of Alberta, Edmonton, Alberta, Canada
- France (4):
  - CHU Toulouse, Toulouse, Haute-Garonne
  - CHRU Nancy Hôpital des Enfants, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Hôpital Necker - Enfants Malades, Paris, Paris
  - CHU de Marseille - Hôpital de la Timone, Marseille
- Italy (3):
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - ASST di Monza - Azienda Ospedaliera San Gerardo, Monza, Monza A Brianza
  - Azienda Ospedaliero Universitaria A Meyer - INCIPIT - PIN, Florence, Tuscany
- Japan (2):
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - The Jikei University School of Medicine, Minato, Tokyo
- Erasmus MC, Rotterdam, South Holland, Netherlands
- Spain (7):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Cruces, Barakaldo
  - Hospital Universitario Raymon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Universitari I Politecnic La Fe de Valencia, Valencia
- United Kingdom (4):
  - Victoria Hospital, Kirkcaldy, Fife
  - St Mary's Hospital - PPDS, Manchester, Lancashire
  - Great Ormond Street Hospital, City of London, London
  - University Hospital Birmingham, Birmingham